CLINICAL TRIAL: NCT03481673
Title: COPE for Children With Asthma: A Cognitive Behavior Skills-Building
Brief Title: COPE for Children With Asthma: Intervention for Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Nurses Foundation (Other); Sigma Theta Tau International Honor Society of Nursing (Other); National Association of Pediatric Nurse Practitioners (Unknown); Sigma Theta Tau Epsilon Branch (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017B0094
Record Dates: First submitted 2017-11-20; First posted 2018-03-29 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Childhood Asthma; Childhood Anxiety Disorder; Childhood Depression
Keywords: Childhood Asthma; Childhood Anxiety; Childhood Depression; Childhood Quality of Life

STUDY DESIGN:
Intervention Model Description: Single group, pre-experimental, intervention pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This pre-experimental pilot project is a single group, pretest-posttest design with a 6-week post-intervention follow-up. A single group design was chosen for this feasibility pilot study because the COPE for Asthma intervention is newly adapted for 8 to 12-year-old children with asthma in an urban setting. The intervention will consist of 7 weekly sessions (30 minutes each). COPE for Asthma is a manualized, cognitive behavior skills-building intervention to improve the physical and mental health outcomes of children with asthma and elevated symptoms of anxiety or depression. Surveys with children and their parents/caregivers (CGs) will occur at baseline, immediately post-intervention and 6 weeks' post-intervention.
  Interventions: Behavioral: COPE for Asthma

INTERVENTIONS:
Behavioral: COPE for Asthma — The intervention will consist of 7 weekly sessions (30 minutes each). COPE for Asthma is a manualized, cognitive behavior skills-building intervention to improve the physical and mental health outcomes of children with asthma and elevated symptoms of anxiety or depression.

SUMMARY:
Children with a chronic condition are at a significantly higher risk for anxiety and depression than those without a chronic condition. Asthma is the most common childhood chronic condition. Children with asthma and co-morbid anxiety and/or depression are at risk of poor health outcomes. The purpose of this study is to evaluate the effects of a manualized cognitive behavior skills-building intervention on key physical and mental health outcomes in 8 to 12-year old children with persistent asthma and co-morbid anxiety and/or depression. The results of this study will inform a large scale randomized controlled trial to fully test this needed intervention.

COPE (Creating Opportunities for Personal Empowerment), developed by Dr. Melnyk, is a manualized intervention that has been implemented with children, adolescents, and young adults. COPE is a cognitive behavior skills-building program based on cognitive behavior theory. Results from previous studies using COPE have shown consistent decreases in anxiety and depression as well as an increase in healthy lifestyle behaviors in youth with elevated anxiety and depressive symptoms in inner city and rural settings, youth with obesity, and teens experiencing chronic recurrent headaches. However, the COPE program has never been adapted and tested with children who have persistent asthma. This study proposes to test an adaptation of this evidence-based program, "COPE for Asthma," with 8 to 12-year-old children with persistent asthma and elevated anxiety and/or depressive symptoms. COPE for Asthma combines components of asthma education with cognitive behavioral skills. This novel adaptation could fill a gap in research by providing a scalable intervention for this highly vulnerable population.

DETAILED DESCRIPTION:
The Interventionist was trained on the implementation of the COPE intervention and will deliver the COPE for Asthma intervention. The intervention, delivered by Colleen McGovern -the Interventionist, will take place in a room within the school separate from other students. The room will include a door for privacy. The intervention will be once/week, 30 minute sessions, for 7 weeks - during lunch and/or recess time. Groups during lunch and recess, or "lunch bunch" groups, are routinely held in the school system by the social workers, guidance counselors, and school nurses. Participants will be given weekly tickets allowing them to get in line first to pick up their lunch to maximize the allotted time. If the material for a session is not covered (i.e., school-wide fire drill, lock down, or other unforeseen event), the session will be moved to the following week.

In the event a participant has severely elevated t-scores, >=70, on the anxiety or depression screening tools or expresses feelings or intent to harm self or others (at any time point or otherwise), the principal, school nurse and/or guidance counselor/social worker will be notified for follow-up per the school district's protocol. A form letter will be sent to the child's CG that day. If child discloses accounts of abuse or neglect, Franklin County Children's Services will be notified and the principal, school nurse and/or guidance counselor/social worker.

Consent/assent of the CG and child and initial screening for anxiety/depression:SCARED and PROMIS measures; will be completed by the Interventionist and a research assistant, RA, from Dr. Melnyk's research team. Data collection and the intervention will start when >=5 child/CG dyads have been consented/assented in a school.

Week 1 at baseline. To avoid bias, the Interventionist will serve as the interventionist and the RA will complete the data gathering. The measures for the child participants will be explained, then self-administered, and checked for completeness by the RA. The RA will conduct phone interviews with the CGs to gather data on demographics, controller medication adherence, and the Asthma Control Test. If phone contact is not possible, the surveys will be sent home with the child with sealable envelopes for the return.

Weeks 2 - 8. COPE for Asthma will be delivered in small groups (Interventionist may need to implement the intervention at several schools on different days; this is expected). Lessons include 30 minutes of didactic teaching and activities.

Post-Intervention Assessment, after the 7-week intervention. After the last COPE for Asthma session has been implemented in a group, a member of Dr. Melnyk's research team will administer the post-intervention follow-up surveys. CGs will be contacted to complete the parent/CG survey.

6-Week Post-Intervention Assessment. The same procedure as for the post-intervention assessment will be conducted for this time period for the children and CGs.

ELIGIBILITY:
Inclusion Criteria:

* Children age 8-12 years enrolled in Columbus City Schools
* Diagnosis of persistent asthma requiring daily inhaled controller medication use at some point (medical condition form on file with the school/CG report)
* Have symptoms depression or anxiety per the PROMIS/SCARED measures
* Have written consent to participate provided by care giver and child assent
* The participating care giver has primary or at least equal responsibility for the day-to-day management of the child's asthma
* care givers provide written consent for their own participation
* Be able to speak, read, and write in English (care giver and child).

Exclusion Criteria:

* has other significant pulmonary conditions (e.g., pulmonary fibrosis, cystic fibrosis)
* currently receiving treatment from a mental health professional
* child or CG has cognitive learning disability that could interfere with the ability to comprehend the interview questions.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Measure change in perception of asthma self-management over three time points | Baseline (week 1, before the intervention starts), post-intervention (week 8-9, after the 7-week intervention), and 6-weeks post-intervention (week 16-17).
  Asthma Management Self-Efficacy: The Child ASE scale (14 items) measures children's perception of their own ability to manage asthma (e.g., "...can tell when a serious breathing problem can be controlled at home"); assesses asthma symptoms, health status, and impact of the child's illness on the family. Higher scores indicate greater self-efficacy; (α=.87). This measure has been validated in children ages 7 - 15 years.

SECONDARY OUTCOMES:
Measure change in anxiety symptoms over three time points | Baseline (before the intervention starts), post-intervention (after the 7-week intervention), and 6-weeks post-intervention.
  Anxiety Symptoms: SCARED (Screen for Child Anxiety Related Emotional Disorders) assesses five factors including panic/somatic, general anxiety disorder, separation anxiety, social phobia, and school phobia; it has been validated with children and adolescents ages 8 - 19 years. Items are scored from 0 (not true or hardly ever true) to 2 (very true or often true). Higher scores indicate greater anxiety with a total score of 25 as having a potential anxiety disorder and 30 as more specific (α=.70 - .90).
Measure change in depressive symptoms over three time points | Baseline (before the intervention starts), post-intervention (after the 7-week intervention), and 6-weeks post-intervention.
  Depressive Symptoms: PROMIS Pediatric Short Form: Assesses negative mood (e.g., sadness), decrease in positive affect (e.g., loss of interest), negative views of self (e.g., worthlessness), and negative social cognition (e.g., loneliness, interpersonal alienation). Items are scored from 0 (never) to 4 (almost always). Higher scores indicate greater anxiety(α=.85). The PROMIS Pediatric Instruments are intended for children between the ages of 8 - 17 years.
Measure change in confidence in managing stress over three time points | Baseline (before the intervention starts), post-intervention (after the 7-week intervention), and 6-weeks post-intervention.
  Personal Beliefs Scale: Child Version: 10-item Likert-type scale with items scored from 1 (strongly disagree) to 5 (strongly agree); assesses personal beliefs and confidence about managing stress. Higher scores indicate greater beliefs (α=.85). This scale has been used in prior studies for children and youth between the ages of 9 - 18 years.
Measure change in symptom interpretation over three time points | Baseline (before the intervention starts), post-intervention (after the 7-week intervention), and 6-weeks post-intervention.
  Symptom Interpretation: Childhood Asthma Symptom Checklist (CASCL): Interpretation of symptoms; 20-item measure of the frequency that children experience physical symptoms, irritability, and panic-fear during asthma attacks.191 Items are scored on a 4-point scale from 1 (never) to 4 (always). In addition to the three subscales the instrument yields a total symptom score (α=.81). This measure has been validated for children between the ages of 6 - 18 years.
Measure change in barriers to controller medications over three time points | Baseline (before the intervention starts), post-intervention (after the 7-week intervention), and 6-weeks post-intervention.
  Asthma Illness Representation Scale (AIRS-C): Child Version: The 17-item AIRS Child (AIRS-C) was designed to identify barriers and risk factors for under-utilization of controller medications. Higher scores indicate closer alignment with the professional model for asthma management. This scale has been adapted from the validated parent version and was tested in a small pilot study with acceptable reliability(α=.84). It has been validated for children between the ages of 6 - 17 years.
Measure change in quality of life over three time points | Baseline (before the intervention starts), post-intervention (after the 7-week intervention), and 6-weeks post-intervention.
  Pediatric Asthma Quality of Life Questionnaire (PAQLQ): 14-item Likert-type scale validated for children between ages 7 - 17 years; measures the functional problems (symptoms, activity limitations, emotional function) that are troublesome to children with asthma.31 Items are scored from 1 (extremely bothered) to 7 (not bothered at all) and the total score is the mean of items. Higher scores denote better QoL.
Measure change in asthma control over three time points | Baseline (before the intervention starts), post-intervention (after the 7-week intervention), and 6-weeks post-intervention.
  Asthma control: The Childhood Asthma Control Test (C-ACT) consists of questions for children (ages 4-11 years; 4 items) and parents (3 items) and the ACT (for individuals 12 years and older) has similar questions which are self-administered. This instruments assesses interference with activities, asthma symptoms, and nighttime awakenings. The C-ACT (α=.79) exhibits good reliability and validity, and classifies children as very poorly controlled, not well-controlled, or well controlled.
Measure comprehension over each lesson | Baseline (before the intervention starts), post-intervention (after the 7-week intervention), and 6-weeks post-intervention.
  Education Manipulation Checks: 4 (ordinal) questions will be asked after each session to evaluate children's comprehension of session content. Answering 3 out of 4 questions correctly indicates understanding. The Interventionist will review the incorrect questions and provide re-education for that item. These questions are age appropriate questions in line with the manual.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen McGovern, PhD(c), Principal Investigator — Ohio State University
Locations (1):
- Columbus City Schools, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akinbami LJ, Simon AE, Rossen LM. Changing Trends in Asthma Prevalence Among Children. Pediatrics. 2016 Jan;137(1):1-7. doi: 10.1542/peds.2015-2354. Epub 2015 Dec 28. PMID 26712860
- [Background] 2. Centers for Disease Control and Prevention. Healthy Schools; asthma and schools. 2015. Retrieved on 3-28-2016 from http://www.cdc.gov/healthyschools/asthma/index.htm
- [Background] 3. American Lung Association. Asthma and Children Fact Sheet. Retrieved on 4-1-2016 from http://www.lung.org/lung-health-and-diseases/lung-disease-lookup/asthma/learn-about-asthma/asthma-children-facts-sheet.html
- [Background] Goodwin RD, Hottinger K, Pena L, Chacko A, Feldman J, Wamboldt MZ, Hoven C. Asthma and mental health among youth in high-risk service settings. J Asthma. 2014 Aug;51(6):639-44. doi: 10.3109/02770903.2014.897728. Epub 2014 Mar 18. PMID 24628526
- [Background] Lu Y, Mak KK, van Bever HP, Ng TP, Mak A, Ho RC. Prevalence of anxiety and depressive symptoms in adolescents with asthma: a meta-analysis and meta-regression. Pediatr Allergy Immunol. 2012 Dec;23(8):707-15. doi: 10.1111/pai.12000. Epub 2012 Sep 9. PMID 22957535
- [Background] Strunk RC, Mrazek DA, Fuhrmann GS, LaBrecque JF. Physiologic and psychological characteristics associated with deaths due to asthma in childhood. A case-controlled study. JAMA. 1985 Sep 6;254(9):1193-8. PMID 4021061
- [Background] Feldman JM, Ortega AN, McQuaid EL, Canino G. Comorbidity between asthma attacks and internalizing disorders among Puerto Rican children at one-year follow-up. Psychosomatics. 2006 Jul-Aug;47(4):333-9. doi: 10.1176/appi.psy.47.4.333. PMID 16844893
- [Background] Goodwin RD, Robinson M, Sly PD, McKeague IW, Susser ES, Zubrick SR, Stanley FJ, Mattes E. Severity and persistence of asthma and mental health: a birth cohort study. Psychol Med. 2013 Jun;43(6):1313-22. doi: 10.1017/S0033291712001754. Epub 2012 Aug 29. PMID 23171853
- [Background] Feldman JM, Siddique MI, Morales E, Kaminski B, Lu SE, Lehrer PM. Psychiatric disorders and asthma outcomes among high-risk inner-city patients. Psychosom Med. 2005 Nov-Dec;67(6):989-96. doi: 10.1097/01.psy.0000188556.97979.13. PMID 16314605
- [Background] Al Aloola NA, Naik-Panvelkar P, Nissen L, Saini B. Asthma interventions in primary schools--a review. J Asthma. 2014 Oct;51(8):779-98. doi: 10.3109/02770903.2014.914534. Epub 2014 May 19. PMID 24730772
- [Background] Yorke J, Fleming SL, Shuldham C. A systematic review of psychological interventions for children with asthma. Pediatr Pulmonol. 2007 Feb;42(2):114-24. doi: 10.1002/ppul.20464. PMID 17186533
- [Background] Ritz T, Meuret AE, Trueba AF, Fritzsche A, von Leupoldt A. Psychosocial factors and behavioral medicine interventions in asthma. J Consult Clin Psychol. 2013 Apr;81(2):231-50. doi: 10.1037/a0030187. Epub 2012 Oct 1. PMID 23025250
- [Background] Shanahan L, Copeland WE, Worthman CM, Angold A, Costello EJ. Children with both asthma and depression are at risk for heightened inflammation. J Pediatr. 2013 Nov;163(5):1443-7. doi: 10.1016/j.jpeds.2013.06.046. Epub 2013 Aug 3. PMID 23919906
- [Background] Goodwin RD, Bandiera FC, Steinberg D, Ortega AN, Feldman JM. Asthma and mental health among youth: etiology, current knowledge and future directions. Expert Rev Respir Med. 2012 Aug;6(4):397-406. doi: 10.1586/ers.12.34. PMID 22971065
- [Background] Feldman JM, Kutner H, Matte L, Lupkin M, Steinberg D, Sidora-Arcoleo K, Serebrisky D, Warman K. Prediction of peak flow values followed by feedback improves perception of lung function and adherence to inhaled corticosteroids in children with asthma. Thorax. 2012 Dec;67(12):1040-5. doi: 10.1136/thoraxjnl-2012-201789. PMID 23154987
- [Background] Melnyk BM, Small L, Morrison-Beedy D, Strasser A, Spath L, Kreipe R, Crean H, Jacobson D, Kelly S, O'Haver J. The COPE Healthy Lifestyles TEEN program: feasibility, preliminary efficacy, & lessons learned from an after school group intervention with overweight adolescents. J Pediatr Health Care. 2007 Sep-Oct;21(5):315-22. doi: 10.1016/j.pedhc.2007.02.009. PMID 17825729
- [Background] Hoying J, Melnyk BM. COPE: A Pilot Study With Urban-Dwelling Minority Sixth-Grade Youth to Improve Physical Activity and Mental Health Outcomes. J Sch Nurs. 2016 Oct;32(5):347-56. doi: 10.1177/1059840516635713. Epub 2016 Mar 29. PMID 27026664
- [Background] Melnyk BM, Jacobson D, Kelly S, Belyea M, Shaibi G, Small L, O'Haver J, Marsiglia FF. Promoting healthy lifestyles in high school adolescents: a randomized controlled trial. Am J Prev Med. 2013 Oct;45(4):407-15. doi: 10.1016/j.amepre.2013.05.013. PMID 24050416
- [Background] Melnyk BM, Kelly S, Jacobson D, Belyea M, Shaibi G, Small L, O'Haver J, Marsiglia FF. The COPE healthy lifestyles TEEN randomized controlled trial with culturally diverse high school adolescents: baseline characteristics and methods. Contemp Clin Trials. 2013 Sep;36(1):41-53. doi: 10.1016/j.cct.2013.05.013. Epub 2013 Jun 5. PMID 23748156
- [Background] Hoying J, Melnyk BM, Arcoleo K. Effects of the COPE Cognitive Behavioral Skills Building TEEN Program on the Healthy Lifestyle Behaviors and Mental Health of Appalachian Early Adolescents. J Pediatr Health Care. 2016 Jan-Feb;30(1):65-72. doi: 10.1016/j.pedhc.2015.02.005. Epub 2015 Apr 10. PMID 25864433
- [Background] Kozlowski JL, Lusk P, Melnyk BM. Pediatric Nurse Practitioner Management of Child Anxiety in a Rural Primary Care Clinic With the Evidence-Based COPE Program. J Pediatr Health Care. 2015 May-Jun;29(3):274-82. doi: 10.1016/j.pedhc.2015.01.009. Epub 2015 Mar 20. PMID 25801377
- [Background] Militello LK, Melnyk BM, Hekler E, Small L, Jacobson D. Correlates of Healthy Lifestyle Beliefs and Behaviors in Parents of Overweight or Obese Preschool Children Before and After a Cognitive Behavioral Therapy Intervention With Text Messaging. J Pediatr Health Care. 2016 May-Jun;30(3):252-60. doi: 10.1016/j.pedhc.2015.08.002. Epub 2015 Oct 1. PMID 26429638
- [Background] Small L, Bonds-McClain D, Melnyk B, Vaughan L, Gannon AM. The preliminary effects of a primary care-based randomized treatment trial with overweight and obese young children and their parents. J Pediatr Health Care. 2014 May-Jun;28(3):198-207. doi: 10.1016/j.pedhc.2013.01.003. Epub 2013 Mar 17. PMID 23511090
- [Background] Hickman C, Jacobson D, Melnyk BM. Randomized controlled trial of the acceptability, feasibility, and preliminary effects of a cognitive behavioral skills building intervention in adolescents with chronic daily headaches: a pilot study. J Pediatr Health Care. 2015 Jan-Feb;29(1):5-16. doi: 10.1016/j.pedhc.2014.05.001. Epub 2014 Jul 10. PMID 25017938
- [Background] Melnyk BM, Jacobson D, Kelly S, O'Haver J, Small L, Mays MZ. Improving the mental health, healthy lifestyle choices, and physical health of Hispanic adolescents: a randomized controlled pilot study. J Sch Health. 2009 Dec;79(12):575-84. doi: 10.1111/j.1746-1561.2009.00451.x. PMID 19909421
- [Background] 26. Franklin County Public Health. Franklin County HealthMap2016. Retrieved on May 10, 2016 from http://www.myfcph.org/pdfs/hstat_FCHealthMap16.pdf
- [Background] Bursch B, Schwankovsky L, Gilbert J, Zeiger R. Construction and validation of four childhood asthma self-management scales: parent barriers, child and parent self-efficacy, and parent belief in treatment efficacy. J Asthma. 1999;36(1):115-28. doi: 10.3109/02770909909065155. PMID 10077141
- [Background] 28. Assessment Center. PROMIS Scoring Manuals. Retrieved on May 10, 2016 from https://www.assessmentcenter.net/Manuals.aspx
- [Background] Fritz GK, Overholser JC. Patterns of response to childhood asthma. Psychosom Med. 1989 May-Jun;51(3):347-55. doi: 10.1097/00006842-198905000-00009. PMID 2734427
- [Background] Sidora-Arcoleo KJ, Feldman J, Serebrisky D, Spray A. Validation of the Asthma Illness Representation Scale-Spanish (AIRS-S). J Asthma. 2010 May;47(4):417-21. doi: 10.3109/02770901003702832. PMID 20528596
- [Background] Juniper EF, Guyatt GH, Ferrie PJ, Griffith LE. Measuring quality of life in asthma. Am Rev Respir Dis. 1993 Apr;147(4):832-8. doi: 10.1164/ajrccm/147.4.832. PMID 8466117
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] Liu AH, Zeiger RS, Sorkness CA, Ostrom NK, Chipps BE, Rosa K, Watson ME, Kaplan MS, Meurer JR, Mahr TA, Blaiss MS, Piault-Louis E, McDonald J. The Childhood Asthma Control Test: retrospective determination and clinical validation of a cut point to identify children with very poorly controlled asthma. J Allergy Clin Immunol. 2010 Aug;126(2):267-73, 273.e1. doi: 10.1016/j.jaci.2010.05.031. Epub 2010 Jul 10. PMID 20624640
- [Background] 34. Muthén L, Muthén B. Mplus user's guide. 1998-2012. Los Angeles, CA.
- [Background] Murphy JM, Bergmann P, Chiang C, Sturner R, Howard B, Abel MR, Jellinek M. The PSC-17: Subscale Scores, Reliability, and Factor Structure in a New National Sample. Pediatrics. 2016 Sep;138(3):e20160038. doi: 10.1542/peds.2016-0038. Epub 2016 Aug 12. PMID 27519444
- [Background] 36. Wang M, Bodner TE. Growth Mixture Modeling Identifying and Predicting Unobserved Subpopulations With Longitudinal Data. Organizational Research Methods. 2007;10(4):635-656.
- [Background] Jacobson D, Melnyk BM. A primary care healthy choices intervention program for overweight and obese school-age children and their parents. J Pediatr Health Care. 2012 Mar;26(2):126-38. doi: 10.1016/j.pedhc.2010.07.004. Epub 2010 Aug 21. PMID 22360932
- [Background] Sidora-Arcoleo K, Feldman J, Serebrisky D, Spray A. Validation of the Asthma Illness Representation Scale (AIRS). J Asthma. 2010 Feb;47(1):33-40. doi: 10.3109/02770900903362668. PMID 20100018
- [Background] Beidas RS, Stewart RE, Walsh L, Lucas S, Downey MM, Jackson K, Fernandez T, Mandell DS. Free, brief, and validated: Standardized instruments for low-resource mental health settings. Cogn Behav Pract. 2015 Feb 1;22(1):5-19. doi: 10.1016/j.cbpra.2014.02.002. PMID 25642130
- [Background] Hale WW 3rd, Crocetti E, Raaijmakers QA, Meeus WH. A meta-analysis of the cross-cultural psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED). J Child Psychol Psychiatry. 2011 Jan;52(1):80-90. doi: 10.1111/j.1469-7610.2010.02285.x. PMID 20662993
- [Background] Birmaher B, Brent DA, Chiappetta L, Bridge J, Monga S, Baugher M. Psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED): a replication study. J Am Acad Child Adolesc Psychiatry. 1999 Oct;38(10):1230-6. doi: 10.1097/00004583-199910000-00011. PMID 10517055
- [Derived] McGovern CM, Hutson E, Arcoleo K, Melnyk B. Considerations in pediatric intervention research: Lessons learned from two pediatric pilot studies. J Pediatr Nurs. 2022 Mar-Apr;63:78-83. doi: 10.1016/j.pedn.2021.10.016. Epub 2021 Nov 1. PMID 34736820